CLINICAL TRIAL: NCT04379219
Title: Surgery Alone Versus Methotrexate Before Surgery in Cases of First Trimester Cesarean Scar Pregnancy: a Randomized Controlled Trial
Brief Title: Surgery Alone Versus Methotrexate Before Surgery in Cesarean Scar Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Maher elesawi kamel elesawi, Lecturer of obstetric and gynecology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.19.10.639.R1.R2.R3
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Cesarean Scar Pregnancy
Keywords: cesarean scar pregnancy, methotrexate, miscarriage, ectopic pregnancy
MeSH Terms: conditions — Abortion, Spontaneous; Pregnancy, Ectopic | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery (Active Comparator): * Valid consent
  * Anathesia , (regional may br converted into general ). IV antibiotic ( cefotaxime 1 gm I.V )
  * Laparotomy transverse incision (pfannenstiel incision)
  * Exploration of the abdominal cavity
  * Identification of the uterus, dissection of the bladder, incision of the uterus and excision of the CSP mass.
  * Surgical repair of the uterine incision, and the abdomen
  Interventions: Drug: Methotrexate
- methotrexate before surgery (Active Comparator): Valid consent
  * patient will receive 50 mgm /m2 of methtrexate after full investigation ( CBC, serum creatinie, AlT, AST), 1 week before surgery.
  * Anathesia , (regional may br converted into general ). IV antibiotic ( cefotaxime 1 gm I.V )
  * Laparotomy transverse incision (pfannenstiel incision)
  * Exploration of the abdominal cavity
  * Identification of the uterus, dissection of the bladder, incision of the uterus and excision of the CSP mass.
  * Surgical repair of the uterine incision, and the abdomen
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — giving methotrexate at least 1 w week before surgery
  Other Names: unitrexate

SUMMARY:
There are no universal treatment guidelines available. The ultimate purpose of the management of CSP is to simultaneously remove the pregnancy and successfully preserve the woman's fertility (Gonzalez & Tulandi, 2017). A variety of medical and surgical treatment modalities for CSP have been reported; however, most of these are based on low-level evidence(Sun et al., 2019).

DETAILED DESCRIPTION:
This will be a randomized clinical trial to evaluate the effect of administration of methotrexate before surgery in reducing bleeding, injury to bladder and ureter, operative time and removing of CSP mass.This will be in comparison to surgery alone in cases of first trimester cesarean scar pregnancy

ELIGIBILITY:
Inclusion Criteria:•

* Gestational age before 13 w
* Past history of 1 or more CS
* Presence of GS implanted on cesareans scar

Exclusion Criteria:

* Presence of severe vaginal bleeding (emergency)
* Previous history of uterine surgery other than CS
* The whole mass is interior and the bulge is more in the cavity
* Bleeding disorder
* Patient not candidate for methotrexate (Positive fetal heart pulsation,
* Patient refuse to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Estimated blood loss intraoperative | intraoperative blood loss
  the amount of blood in soaked towels and vacuum aspiration

SECONDARY OUTCOMES:
need further management | 1 month
• Rate of urological injury | immediatly and 1 week post operative
• Rate of readmission, relaparotomy | with in 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Maher Elgaly, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes